CLINICAL TRIAL: NCT05272917
Title: SOMESThesia in Patients With Head and Neck Cancer: Variability and Influence on the ALIMentation Experience
Brief Title: SOMESThesia and ALIMentation
Acronym: SOMEST'ALIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL21_1153
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancers
Keywords: Head and Neck cancers; nutrition; somesthesia
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- head and neck cancer patients with radiotherapy AND chemotherapy (Experimental): patients included for a head and neck cancer and treated by radiotherapy (+/- surgery) + chemotherapy
  Interventions: Other: Sensorial tests; Behavioral: food preferences questionnaires
- head and neck cancer patients with radiotherapy only (Experimental): patients included for a head and neck cancer and treated by radiotherapy (+/- surgery) without chemotherapy
  Interventions: Other: Sensorial tests; Behavioral: food preferences questionnaires
- healthy volunteers (Active Comparator): healthy volunteers paired with experimental patients on age (+/- 5 years), gender, tobacco status
  Interventions: Other: Sensorial tests; Behavioral: food preferences questionnaires

INTERVENTIONS:
Other: Sensorial tests — Patients will be included in the study between 3 to 6 months after the end of treatment and go to the Paul Bocuse Research Institute to perform several sensorial tests. The same sensorial tests will be completed by healthy volunteers to compare.
Behavioral: food preferences questionnaires — Patients will be included in the study between 3 to 6 months after the end of treatment and go at Institut Paul Bocuse to complete food preferences questionnaires. The same questionnaires will be completed by healthy volunteers to compare.

SUMMARY:
Cancer patients are at high risk for undernutrition. A study with head and neck cancer patients showed that 50% suffered from undernutrition (Prevost et al., 2014). Sensory alterations may also involve sensory changes from the physiological structures of the mouth or neural pathways and hedonic changes, i.e., although food may taste the same as usual, that taste is no longer judged as pleasant. These changes lead to an aversion to food and a decrease in the pleasure of eating (Bernhardson et al., 2009).

Despite the large number of published studies on taste and smell alterations in diverse cancer populations, few have examined other dimensions of oral sensory alterations. Studies focusing on somesthesia have mostly been conducted in the area of oral physiology or stomatology in relation to oral pain and rehabilitation (Howes, Wongsriruksa, Laughlin, Witchel, & Miodownik, 2014).

Regarding food perception, somesthesia provides information about both texture, temperature, and trigeminal sensations. These sensations are detected by mechanical, thermal, nociceptive receptors present throughout the oral epithelium (Simons & Carstens, 2008). In addition to taste and smell, food perception is influenced by oral somatosensation and studies have demonstrated an interrelated relationship between these oral sensations (Spence, Piqueras-Fiszman 2016). Therefore, ther might have a correlation between oral somatosensation and food preferences, subsequently influencing eating behavior and food consumption. A standard method, using a so-called Von Frey Hair monofilament, to assess tactile sensation was developed by Etter et al. (Etter, N. M et al.,. J. Vis. Exp. 2020) but has so far been only minimally used in Ear, Nose and Throat (ENT) cancer (Bearelly, Wang, & Cheung, 2017; Bodin, Jäghagen, & Isberg, 2004; Elfring, Boliek, Seikaly, Harris, & Rieger, 2012).

The aim of the study is to determine the variability and role of somatosensory perception (texture, pungency transmitted through the trigeminal system, and temperature) on food preferences in cancer patients compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Person between 18 and 65 years
* Person having given free, informed, express written consent
* Person affiliated to a French social security system
* Person with a body mass superior to 18 kg/m².
* Person able to come once to the Institut Paul Bocuse

Patients with head and neck cancer with chemotherapy:

- Patient diagnosed with squamous cell head and neck cancer with the following treatment regimen: Surgery + radiochemotherapy or radiochemotherapy alone

Patients with head and neck cancer without chemotherapy:

- Patient diagnosed with squamous cell head and neck cancer with the following treatment regimen: Surgery + radiation therapy or radiation therapy alone

Healthy volunteers :

* Volunteer who is +/- 5 years of age relative to the patient to whom they are matched.
* Volunteer of the same sex as the patient to whom they are matched
* Volunteer with the same smoking status as the patient to whom they are matched
* Volunteer who has not had cancer within 5 years at the time of inclusion
* Volunteer with no current treatment that may affect taste and smell perception

Exclusion Criteria:

All subjects:

* Person with a known food allergy/intolerance (lactose or milk protein) or unable to consume dairy or solid products (e.g., chocolate milk pudding, chocolate jelly)
* Person with a known allergy to chili (or capsaicin)
* Person with diagnosed total ageusia
* Person with diagnosed total anosmia
* Person who has used artificial feeding within 2 months prior to inclusion.
* Person who has lost more than 10% of baseline weight in the 2 months prior to inclusion
* Person deprived of liberty or under guardianship or trusteeship.
* Pregnant or breastfeeding woman
* Person deprived of liberty by a judicial or administrative decision
* Person under guardianship or protection of vulnerable adults
* Person with trismus (reduced jaw opening or limited jaw range of motion)
* A person who is unable to extend his or her tongue
* Person who has had surgery on the mobile tongue and/or base of the tongue
* Person unable to swallow soft foods
* Person who has had or is suspected of having had Corona Virus Disease (COVID)-19 within the last 6 months.

Patients with head and neck cancer:

* Patient receiving immunotherapy
* Patient treated with surgery only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Oral tactile sensitivity score | Up to 3 months after recruitment.
  The primary endpoint of the study is to measure oral tactile sensitivity using the Von Frey Hair monofilament pressure test in head and neck cancer patients compared to healthy volunteers. This will be assessed at recruitment for healthy volunteers and between 1 to 3 months after recruitment for head and neck cancer patients.

SECONDARY OUTCOMES:
thermic sensitivity score | Up to 3 months after recruitment.
  Measurement on a visual analog scale (gLMS) of sensitivity to heat and cold using dental mirrors. This will be assessed at recruitment for healthy volunteers and between 1 to 3 months after recruitment for head and neck cancer patients.
trigeminal sensitivity score | Up to 3 months after inclusion.
  Visual analog scale (gLMS) measurement of trigeminal sensitivity using prepared solutions. This will be assessed at inclusion for healthy volunteers and between 1 to 3 months after inclusion for head and neck cancer patients.
texture sensitivity score | Up to 3 months after recruitment.
  Measurement of texture sensitivity (firmness, consistency, and roughness) on a visual analog scale (gLMS) from food samples. This will be assessed at recruitment for healthy volunteers and between 1 to 3 months after recruitment for head and neck cancer patients.
salivary function | Up to 3 months after recruitment.
  Saliva function measurement with a BUFFER Saliva-check kit. This will be assessed at recruitment for healthy volunteers and between 1 to 3 months after recruitment for head and neck cancer patients.
food preference score | Up to 3 months after recruitment.
  Measurement of food preference based on food pictures on a visual analog scale and according to the participant's ethnicity, family and social status. This will be assessed at recruitment for healthy volunteers and between 1 to 3 months after recruitment for head and neck cancer patients.
sensory perception, dietary habits and oral health | Up to 3 months after recruitment.
  Measured by self-reported questionnaires of subjective sensory perception, dietary habits, and oral health and according to the participant's ethnicity, family and social status. This will be assessed at recruitment for healthy volunteers and between 1 to 3 months after recruitment for head and neck cancer patients.
correlation sensory perception and food preferences | Up to 3 months after recruitment.
  Correlation analysis between sensory perception and food preferences for each participant. This will be assessed at recruitment for healthy volunteers and between 1 to 3 months after recruitment for head and neck cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Amandine BRUYAS, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Centre de recherche de l'Institut Paul Bocuse, Écully
  - Service d'Oncologie médicale, Hôpital de la Croix-Rousse, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riantiningtyas RR, Valenti A, Dougkas A, Bredie WLP, Kwiecien C, Bruyas A, Giboreau A, Carrouel F. Oral somatosensory alterations and salivary dysfunction in head and neck cancer patients. Support Care Cancer. 2023 Oct 13;31(12):627. doi: 10.1007/s00520-023-08086-7. PMID 37828382